CLINICAL TRIAL: NCT06259227
Title: Personalized Cardiorespiratory Fitness Training in Patients with Incomplete Spinal Cord Injury During Primary Rehabilitation
Brief Title: Cardiorespiratory Fitness Training in Patients with Incomplete Spinal Cord Injury
Acronym: FIT@HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1045; NL81465.091.22 (Other: CCMO)
Record Dates: First submitted 2023-09-18; First posted 2024-02-14 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Incomplete Spinal Cord Injury; Exercise Training
MeSH Terms: interventions — Cardiorespiratory Fitness; Corticotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): During the primary rehabilitation program, the intervention group will receive 2-3 individualized cardiorespiratory fitness training sessions per week.
  Interventions: Other: Cardiorespiratory fitness (CRF) training
- Control group (No Intervention): The control group will receive usual care.

INTERVENTIONS:
Other: Cardiorespiratory fitness (CRF) training — The CRF training will take place on an arm cycle ergometer, or on an recumbent cross trainer. The duration and intensity of these 2 CRF gait training sessions will be determined by scientific exercise guidelines. A practical way of increasing vigorous-intensity exercise is high-intensity interval training (HIIT). The HIIT intervention consist of 2-3 trainings per week, with each exercise session including a 5-minute warm-up, 30-second interval periods (with a power output up to 90% of the peak power output (PPO)), and 30-second recovery periods. There are 5 minutes of 50% of PPO between interval periods. The number of interval periods increases during the intervention period, resulting in a maximum total training time of 35 minutes.
  Arms: Intervention group

SUMMARY:
The goal of this exploratory randomized controlled trial is to assess the effect of a personalized training intervention during primary rehabilitation of 6 weeks on cardiorespiratory fitness in individuals with subacute (<6 months) spinal cord injury during primary rehabilitation and during follow-up. Secondary outcomes include the effect on gait assessments, pulmonary function, neurological status, muscle force, cardiometabolic risk factors, quality of life, functional independence and self-efficacy.

Participants in the intervention group will receive 2-3 personalized cardiorespiratory fitness-focused training sessions per week, for a period of 6 weeks. Participants in the control group will receive usual care.

DETAILED DESCRIPTION:
Rationale:

Despite advances in medical care, spinal cord injury (SCI) patients have significantly lower survival rates compared to the general population. The 'Koepelproject', an unique world-leading multi-center research project, discovered that SCI patients have a decreased pulmonary function, which is linked to poor cardiorespiratory fitness (CRF). This leads to respiratory and cardiovascular diseases, which are important predictors of death in SCI patients. However, there are limitations of the 'Koepelproject' which highlight the need for the proposed project 'FIT@HOME'. Rehabilitation knowledge in SCI patients is primarily focused on those with a complete lesion, while there has been changes in the characteristics of the SCI population over the last few decades. The diagnosis of an incomplete SCI (iSCI) is more common and requires different insights and skills compared to patients with complete lesions. Therefore, insight in the effect of personalized rehabilitation strategies focussed on CRF during primary rehabilitation will provide important information to support healthy ageing in iSCI patients.

Objective:

The primary aim of this study is to assess the effect of a personalized training intervention on CRF during primary rehabilitation and at follow-up. Secondary aims of this study are to determine the effect of this training intervention on gait capacity, pulmonary function, neurological status, muscle force, cardiometabolic risk factors, quality of life (QoL), functional independence and exercise self-efficacy.

Study design:

The proposed study design is an explorative randomized controlled trial.

Study population:

This study will include 32 iSCI patients classified with an American Spinal Injury Association (ASIA) C or D in the subacute phase (< 6 months post injury), who are referred for a primary, inpatient rehabilitation program at the Sint Maartenskliniek.

Intervention:

The intervention includes 2-3 personalized CRF-focused training sessions per week. The control group receives usual care.

Main study parameters/endpoints:

The primary endpoint is the change in CRF (expressed as VO2peak) after the 6-weeks intervention period and at follow-up.

Secondary outcomes are gait assessments, pulmonary function, neurological status, muscle force, cardiometabolic risk factors, secondary complications, quality of life, functional independence and exercise self-efficacy.

Measurements will be performed at:

T0 - Baseline

T1 - Following the 6-weeks intervention period during the primary rehabilitation program at the Sint Maartenskliniek

T2* - At discharge from the primary rehabilitation program at the Sint Maartenskliniek (only if the period following T1 is more than 2 weeks)

T3 - After 2 weeks in the outpatient rehabilitation program at the Sint Maartenskliniek

T4 - At discharge from the outpatient rehabilitation program at the Sint Maartenskliniek

T5 - 2 weeks following discharge from the outpatient rehabilitation program at the Sint Maartenskliniek (2 weeks after T4)

T6 - 3 months following discharge from the outpatient rehabilitation program at the Sint Maartenskliniek (3 months after T4, 2.5 months after T5)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of incomplete spinal cord injury based on a stable cause (e.g. traumatic)
* Spinal cord injury classification C or D on the American Spinal Injury Association (ASIA) impairment scale
* During this study in the subacute phase (< 6 months post injury)
* Hospitalized in the Sint Maartenskliniek for a primary, inpatient rehabilitation program
* Older than 18 years of age
* Able to understand and perform study related procedures
* Capable to sit at least 3 times a day for 2 hours (prerequisites to start the active rehabilitation program)
* The ability to use an arm ergometer

Exclusion Criteria:

* Unable to give informed consent
* Language barrier
* Participating in another interventional study targeting cardiorespiratory fitness
* Have contraindications to perform exercise during the rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Defined as VO2peak in ml/kg/min

SECONDARY OUTCOMES:
Gait assessments - Walking ability | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), 2 weeks after T2 (T3), end of outpatient rehab (T4) (average 3 months after T2) , 2 weeks after T4 (T5), 3 months after end of outpatient rehab (T6)
  Measured by Walking Index of Spinal Cord Injury (WISCI II), which is an ordinal scale (0-20) consisting of 21 items reflecting various levels of walking ability, taking into account the use of assistive devices, orthotic devices and physical assistance.
Gait assessments - Gait capacity | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), 2 weeks after T2 (T3), end of outpatient rehab (T4) (average 3 months after T2) , 2 weeks after T4 (T5), 3 months after end of outpatient rehab (T6)
  Measured by the self-paced 2-Minute-Walk-Test (2MWT). Participants will be instructed to walk as far as possible at a comfortable walking speed in two minutes. The total distance walked in meters will be recorded. Furthermore, participants will be fitted with a facemask that will allow for the collection of respiratory gasses. Oxygen uptake and heart rate will be measured during the 2MWT (walking efficiency).
Gait assessments - Gait performance | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), 2 weeks after T2 (T3), end of outpatient rehab (T4) (average 3 months after T2) , 2 weeks after T4 (T5), 3 months after end of outpatient rehab (T6)
  Daily life gait performance is measured by inertial measurements units (IMU), determining spatiotemporal parameters. Furthermore, the Activ8 activity monitor will be used.
Pulmonary function - Forced Vital Capacity (FVC) | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by simple spirometry and defined as the total volume of air that a person can forcibly exhale during a maximal expiratory effort in liters.
Pulmonary function - Forced Expiratory Volume in 1 second (FEV1) | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by simple spirometry and defined as the volume expired in the first second of the FVC maneuver in liters.
Pulmonary function - Peak Expiratory Flow (PEF) | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by simple spirometry and defined as the maximal expiratory flow rate achieved during the FVC maneuver and is defined in liters/minute.
Neurological status | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by the ASIA impairment scale will be used for both a motor and sensory examination. The ASIA impairment scale consists of a 5-point ordinal scale, which classifies individuals from "A" (complete SCI) to "E" (normal sensory and motor function).
Muscle force - Grip force | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by handgrip strength of the dominant hand. This will be assessed with a hydraulic, analogue hand dynamometer adjusted to the hand size of every participant.
Muscle force - Voluntary muscle strength | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Voluntary muscle strength of 5 key muscles of both lower extremities and key muscles of both upper extremities in accordance with standard neurological assessment (ASIA). A six-point scale is used for scoring with 0 being total paralysis and 5 is normal active moment, full range of motion against gravity and expected from an unimpaired person.Upper extremity muscle strength will also be measured using a handheld dynamometer (HHD).
Cardiometabolic risk factors - Waist circumference (cm) | Baseline (T0) , 3 months after end of outpatient rehab (T6)
  Measured in a standing position across the belly button during the exhale.
Cardiometabolic risk factors - Skinfold thickness | Baseline (T0) , 3 months after end of outpatient rehab (T6)
  Measured by a skinfold calliper and will be performed according to the American College of Sports Medicine standard description of skinfold measurements.
Cardiometabolic risk factors - Blood pressure | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Descriptive outcome measure in mmHg
Cardiometabolic risk factors - Heart rate | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Descriptive outcome measure in beats per minute
Cardiometabolic risk factors - Low Density Lipoprotein Cholesterol (LDL-C) | Baseline (T0) , 3 months after end of outpatient rehab (T6)
  Measured by a venous blood sample when participants have been sober for 4 hours
Cardiometabolic risk factors - High Density Lipoprotein Cholesterol (HDL-C) | Baseline (T0) , 3 months after end of outpatient rehab (T6)
  Measured by a venous blood sample when participants have been sober for 4 hours
Cardiometabolic risk factors - Total Cholesterol (TC) | Baseline (T0) , 3 months after end of outpatient rehab (T6)
  Measured by a venous blood sample when participants have been sober for 4 hours
Cardiometabolic risk factors - Fasted insulin | Baseline (T0) , 3 months after end of outpatient rehab (T6)
  Measured by a venous blood sample when participants have been sober for 4 hours
Cardiometabolic risk factors - Fasted glucose | Baseline (T0) , 3 months after end of outpatient rehab (T6)
  Measured by a venous blood sample when participants have been sober for 4 hours
Secondary complications - Urinary and bowel dysfunction | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Descriptive outcome measure
Secondary complications - Level of pain experienced during the last week | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by the visual analog scale (VAS). The VAS is an unidimensional measure, containing a straight horizontal line of 100 mm. Furthermore, pain will be classified according to the type of pain (neuropathic or nociceptive (musculoskeletal / visceral / other).
Secondary complications - Shoulder pain | Baseline (T0), 6 weeks after T0 (T1)
  Measured by the pain subscale of the Shoulder Pain and Disability Index (SPADI) questionnaire. The subscale consists of five items on the numerical rating scale from 0 to 10, with a higher value indicating more disability.
Secondary complications - Level of fatigue experienced during the last week | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by the visual analog scale (VAS). The VAS is an unidimensional measure, containing a straight horizontal line of 100 mm.
Secondary complications - Pressure sores | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Descriptive outcome measure including location, severity and duration
Secondary complications - Spasticity | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Measured by the Modified Ashworth Scale (MAS). The MAS is a scale of perceived resistance (tone) against passive movement of the limb and is the most widely used scale in the clinical setting. MAS assigns a grade of spasticity from a 0-4 ordinal scale, where lower scores represent normal muscle tone and higher scores represent spasticity.
Secondary complications - Number of respiratory and cardiovascular complications | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Descriptive outcome measure
Secondary complications - Number of rehospitalizations | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Descriptive outcome measure
Quality of Life (QoL) | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), 2 weeks after T2 (T3), end of outpatient rehab (T4) (average 3 months after T2) , 2 weeks after T4 (T5), 3 months after end of outpatient rehab (T6)
  Measured by the Quality of Life Basic Data Set Version 2.0 (QoL-BDS V2.0). This questionnaire includes four items on the individual's satisfaction with their life as a whole, their physical health, mental health, and social life. All items use a 0-10 numerical rating scale with higher scores indicating better QoL.
Functional independence | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), 2 weeks after T2 (T3), end of outpatient rehab (T4) (average 3 months after T2) , 2 weeks after T4 (T5), 3 months after end of outpatient rehab (T6)
  Measured by the Spinal Cord Independence Measure III (SCIM III). This questionnaire includes three specific areas of function: selfcare, respiration and sphincter management and a patient's mobility abilities. Each subscale score is evaluated within the 100-point scale, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence.
Exercise self-efficacy | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), 2 weeks after T2 (T3), end of outpatient rehab (T4) (average 3 months after T2) , 2 weeks after T4 (T5), 3 months after end of outpatient rehab (T6)
  Measured by the exercise self-efficacy scale (ESES). The ESES consists of 10 items about level of self-confidence with regard to performing regular physical activities and exercise.

OTHER OUTCOMES:
Age (years) | Baseline (T0)
  Descriptive outcome measure
Sex (male / female) | Baseline (T0)
  Descriptive outcome measure
Height (cm) | Baseline (T0)
  Descriptive outcome measure
Weight (kg) | Baseline (T0)
  Descriptive outcome measure
Body Mass Index (kg/m^2) | Baseline (T0)
  Descriptive outcome measure
Nationality | Baseline (T0)
  Descriptive outcome measure
Medical history | Baseline (T0)
  Descriptive outcome measure
Time since spinal cord injury (days) | Baseline (T0)
  Descriptive outcome measure
Cause of spinal cord injury (traumatic / non-traumatic) | Baseline (T0)
  Descriptive outcome measure
Level of spinal cord injury | Baseline (T0)
  The level of injury for a person with SCI is the lowest point on the spinal cord below which sensory feeling and motor movement diminish or disappear. The level is denoted by the letter-and-number name of the vertebra at the injury site (such as C3, T2, or L4).
Medication use | Baseline (T0), 6 weeks after T0 (T1), end of inpatient rehab (T2)* (average 3 months after T0), end of outpatient rehab (T4) (average 3 months after T2) , 3 months after end of outpatient rehab (T6)
  Medication that could influence outcome measures (e.g. beta-blockers, antihypertensives, statins).
Smoking history | Baseline (T0)
  Descriptive outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Ilse van Nes, Dr., Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands

IPD SHARING:
Plan to Share IPD: No